CLINICAL TRIAL: NCT06224218
Title: Randomized Controlled Trial Comparing Single Port Simple Prostatectomy and Laser Enucleation of the Prostate for Benign Prostatic Hyperplasia
Brief Title: Prostate Single Port & Laser Enucleation Comparison Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Simone Crivellaro, Urology Dpt, Vice Chair, Lawrence S. Ross Endowed Professor & Associate Professor of Urology Robotic, Section Chief, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 2023-1335
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Port Robotic Prostatectomy (Active Comparator): Removal of the prostate using single port robot
  Interventions: Procedure: Single Port Robotic Surgery
- Laser Enucleation of the Prostate (Active Comparator): Enucleation of the prostate with laser surgery
  Interventions: Procedure: Laser Surgery

INTERVENTIONS:
Procedure: Single Port Robotic Surgery — Single port Robotic surgery will remove the whole prostate
  Arms: Single Port Robotic Prostatectomy
Procedure: Laser Surgery — Laser enucleation will remove chips of the prostate but keeping intact the prostate capsule.
  Arms: Laser Enucleation of the Prostate

SUMMARY:
Surgical treatments for benign prostatic hyperplasia (BPH) are necessary when non-procedural approaches fail to alleviate lower urinary tract symptoms (LUTS) or bladder outlet obstruction (BOO). Open simple prostatectomy and laser enucleation are recommended for prostatic adenoma size greater than 80 ml. Minimally invasive approaches, such as robotic-assisted simple prostatectomy, have gained popularity due to their comparable outcomes with lower morbidity. The introduction of the da Vinci single-port (SP) robotic platform offers potential advantages, but its outcomes have not been thoroughly investigated.

This randomized controlled trial aims to compare the outcomes of SP simple prostatectomy performed using the da Vinci robotic platform versus thulium laser enucleation of the prostate for the treatment of BPH and BOO.

DETAILED DESCRIPTION:
Patients diagnosed with symptomatic BPH and eligible for surgical intervention will be randomized to undergo either SP robotic simple prostatectomy or thulium laser enucleation of the prostate. Primary outcomes will include perioperative parameters (operative time, estimated blood loss, hospital stay), postoperative complications, and functional outcomes (urinary symptoms, urinary flow rate). Secondary outcomes will evaluate perioperative and postoperative complications, oncologic outcomes, and patient-reported quality of life measures.

In a recent retrospective study at UI Health from 2017 to 2021, investigators compared 103 procedures, SP robotic prostatectomy versus laser enucleation, 34 SP robotic prostatectomy and 69 laser enucleations. There was no difference in any complication at 30-day post-surgery (21.2% vs. 21.7%, p=0.9517). Investigators recognize SP robotic surgery leads to longer operating times, due to docking the instrument and closing the incision, as well as longer catheter times to allow the cystostomy to heal. While the laser enucleation may be considered less invasive, as no incision is required, the instrumentation of the urethra could lead to urethral strictures. This study aims to provide valuable insights into the clinical outcomes of single port simple prostatectomy using SP robotic platform, compared to laser enucleation of the prostate prospectively. The results of this trial will help guide clinicians and patients in selecting the most appropriate surgical intervention for symptomatic BPH, considering both functional outcomes and morbidity. Both procedures are currently performed at UI Health, they are FDA approved, therefore this is not a safety study. Subject insurance will not impact which subject will receive one procedure or the other, as both procedures are recommended on the American Urological Association guidelines for Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia.

The study will be a randomized controlled trial comparing SP simple prostatectomy vs laser enucleation of the prostate. The study findings will improve clinical decision-making and aid in optimizing patient outcomes in the management of BPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with symptomatic Benign Prostatic Hyperplasia (BPH) who fail conservative treatment with drug therapy are eligible for surgical intervention.

Exclusion Criteria:

* Adults unable to consent Prisoners Cognitive impaired adults Coagulopathy

Ages: 18 Years to 88 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Operative time | During procedure
  Time in minutes from the start to finish of the procedure.
International Consultation of Incontinence Questionnaire Short Form | Before procedure and 7 months after procedure
  How often do you leak urine? never 0 about once a week 1 two or three times a week 2 about once a day 3 several times a day 4 all the time 5
  How much urine do you usually leak (whether you wear protection or not)? none 0 a small amount 2 a moderate amount 4 a large amount 6
  Overall, how much does leaking urine interfere with your everyday life? 0 (not at all) and 10 (a great deal) 0 1 2 3 4 5 6 7 8 9 10
  ICIQ score: sum previous questions.
  When does urine leak? never - urine does not leak before you can get to the toilet when you cough or sneeze when you are asleep when you are physically active/exercising when you have finished urinating and are dressed for no obvious reason all the time
Sexual Health Inventory for Men (SHIM) | Before procedure and 7 months after procedure
  1. How do you rate your confidence to keep an erection? 1 Very low 2 3 4 5 Very high
  2. How often were your erections hard enough for penetration? 1 Almost never 2 3 4 5Almost always
  3. How often were you able to maintain your erection after you had penetrated your partner? 1Almost never 2 3 4 5Almost always
  4. How difficult was it to maintain your erection to completion of intercourse? 1Extremely difficult 2 3 4 5Not difficult
  5. When you attempted sexual intercourse, how often was it satisfactory for you? 1Almost never 2 3 4 5Almost always
  Add together the numbers. If the patient's score is 21 or less, erectile dysfunction (ED) should be addressed.
  22 - 25: No significant erectile dysfunction 17 - 21: Mild erectile dysfunction 12 - 16: Mild-to-moderate erectile dysfunction 8 - 11: Moderate erectile dysfunction 5 - 7: Severe erectile dysfunction
International Prostate Symptom Score I-PSS | Before procedure and 7 months after procedure
  1. How often have you had a sensation of not emptying your bladder completely after you finish urinating?
  0= not all
  1. less than 1 time in 5
  2. less than half the time
  3. about half the time
  4. more than half the time
  5. almost always
  2. How often have you had to urinate again less than two hours after you have finished urinating?
  0 1 2 3 4 5
  3. How often have you found you stopped and started again several times when you urinated?
  0 1 2 3 4 5
  4. How often have you found it difficult to postpone urination?
  0 1 2 3 4 5
  5. How often have you had a weak urinary stream?
  0 1 2 3 4 5
  6. How often have you had to push or strain to begin urination?
  0 1 2 3 4 5
  7. How many times did you most typically get up each night to urinate from the time you went to bed until the time you got up in the morning?
  0 1 2 3 4 5
  Sum previous questions to have the score:
  0 - 7 = mildly symptomatic; 8 - 19 = moderately 20 - 35 = severely
Urinary flow rate | Before procedure and 7 months after procedure
  Measure of the urine flow in mL/s
Post void residual volume | Before procedure and 7 months after procedure
  Amount of urine retained in the bladder after a voluntary void measure with Ultrasound.
  Volume = length x width x height x 0.52
Blood loss during procedure | During procedure
  Estimate blood loss in mL during procedure
Hospital stay after procedure | From end of procedure to discharge home (up to 30 days )
  Amount of time spent at the hospital after procedure measure in hours

SECONDARY OUTCOMES:
Number of subjects with injuries related to surgical procedures. | During procedure
  Descriptive report of complications during surgery.
Quality of life due to urinary symptoms | Before procedure and 7 months after procedure
  If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?
  0 1 2 3 4 5 6
  0= delighted
  1. please
  2. mostly satisfied
  3. mixed
  4. mostly unhappy
  5. unhappy
  6. terrible
Number of subjects with incidental cancer | 2 weeks after procedure
  Pathology report of prostate tissue, presence or absence of prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Crivellaro, MD, Principal Investigator — University of Illinois at Chicago, Department of Urology
Locations (1):
- UI Health SCB Clinic Department of Urology, Chicago, Illinois, United States

REFERENCES:
- [Result] Talamini S, Lai A, Palmer C, van de Walle G, Zuberek M, Crivellaro S. Surgical treatment of benign prostatic hyperplasia: Thulium enucleation versus single-port transvesical robotic simple prostatectomy. BJUI Compass. 2023 Jun 22;4(5):549-555. doi: 10.1002/bco2.261. eCollection 2023 Sep. PMID 37636211
- [Result] Bove AM, Brassetti A, Ochoa M, Anceschi U, D'Annunzio S, Ferriero M, Tuderti G, Misuraca L, Mastroianni R, Cartolano S, Torregiani G, Lombardo R, De Nunzio C, Simone G. Robotic simple prostatectomy vs HOLEP, a 'multi single-center' experiences comparison. Cent European J Urol. 2023;76(2):128-134. doi: 10.5173/ceju.2023.204. Epub 2023 Apr 17. PMID 37483855